CLINICAL TRIAL: NCT05746195
Title: Use of Text Messages to Increase Whole Grain Consumption in Colorectal Cancer
Brief Title: Optimization of Adaptive Text Messages for Cancer Survivors (OATS II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 224523; NCI-2023-00870 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); R21CA263539 (NIH)
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Colon Adenocarcinoma; Colorectal Carcinoma; Rectal Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Text message intervention (Experimental): Adaptive 12-week text message intervention using reinforcement learning to increase whole grain and reduce refined grain intake via the HealthySMS platform. Participants will also complete semi-structured follow-up interviews and various questionnaires evaluating participants dietary habits and use of study intervention.
  Interventions: Behavioral: Dietary intervention via Text Messaging; Other: Survey Administration; Behavioral: Nutrition Education

INTERVENTIONS:
Behavioral: Dietary intervention via Text Messaging — Text messages will be sent to participants cell phones using the HealthySMS platform
Other: Survey Administration — Various questionnaires evaluating participants dietary habits and use of study intervention will be administered
Behavioral: Nutrition Education — Participants will receive nutrition education materials

SUMMARY:
This clinical trial evaluates whether an adaptive text-message intervention is useful in helping survivors of colorectal cancers (CRC) eat more whole grain foods and less refined grain foods. Most CRC survivors don't achieve the recommended intakes of whole grains or fiber, even though there is strong evidence that a high-fiber diet rich in whole grains lowers the risk of death from CRC. Dietary interventions are a promising approach for reducing death from CRC, and text message interventions specifically are a promising tool for reaching diverse populations. This trial evaluates a text-message based dietary intervention that continuously adapts message content to be specifically tailored for the participant for increasing whole grain consumption.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the intervention's feasibility and acceptability.

SECONDARY OBJECTIVES:

I. Estimate the effect of the intervention on the percent of grains consumed that are whole.

II. Estimate the effect of the intervention on total fiber intake (grams per day [g/d]).

EXPLORATORY OBJECTIVE:

I. Assess convergence of the reinforcement learning (RL) algorithm.

OUTLINE:

Patients receive nutrition education materials and then receive the adaptive text message intervention for 12 weeks on study. Patients who are food insecure also receive resources for food banks, information about meal delivery programs, and support for applying for Supplemental Nutrition Assistance Program (SNAP) benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Subject has provided informed consent.
3. Diagnosis of colon or rectal adenocarcinoma.
4. Not on active treatment at the time of screening and not expected to receive active anticancer therapy (e.g., surgery, radiation, chemotherapy) during the study period.
5. At least 6 weeks since a major surgery and fully recovered.
6. Owns a mobile phone and is willing and able to receive and send text messages.
7. Able to speak/read English or Spanish.
8. Based on a screening survey, eat grains and =<50% of total grains are whole grains.

Exclusion Criteria:

1. Does not meet any of the above inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Van Blarigan, ScD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Zuckerberg San Francisco General, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Text Message Intervention
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Text Message Intervention
Number analyzed (Participants) | 46
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 2
  40-49 years old | 5
  50-59 years old | 12
  60-69 years old | 16
  70-79 years old | 8
  80-89 years old | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 7
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Median Percentage of Text Messages That Participants Responded to That Asked for a Reply
Description: The percentage of text messages responded to is defined as the number of text messages with a response divided by the total number of text messages that ask for a reply and calculated on a per patient basis. The intervention will be determined feasible if the median response rate (percentage of text messages that participants responded to) across all participants is >= 70%.
Time Frame: Up to 12 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of text messages
Arm/Group | Text Message Intervention
Number analyzed (Participants) | 46
percentage of text messages | 96 [90 to 98]

2. Primary Outcome: Overall Median Score on the System Usability Scale (SUS)
Description: The system usability is comprised of 10 questions assessing participants perceived usability of the intervention. Each item is scored on a scale of 1 (strongly disagree) to 5 ( strongly agree). The SUS yields a single number representing a composite measure of the overall usability of the text messaging system. To calculate the SUS score, Each item's score contribution will ultimately range from 0 to 4 (For items 1,3,5,7,and 9 the score contribution is the item score minus 1 and for items 2,4,6,8 and 10, the contribution is the item score minus 5). The sum of the scores are then multiplied by 2.5 to obtain the overall value. SUS scores have a range of 0 to 100 with a score > 68 indicating above average usability.
Time Frame: At 12 weeks
Population: Two participants did not complete this survey at 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Text Message Intervention
Number analyzed (Participants) | 44
score on a scale | 72.5 [65 to 85]

3. Primary Outcome: Overall Score on the Acceptability of Intervention Measure (AIM)
Description: The AIM is a four-item measure of implementation that assesses participants perceived acceptability of the intervention. Each item response falls on a scale of 1 (Completely disagree) to 5 (Completely agree). A scaled score is calculated by averaging responses. Scale values range from 1 to 5. The intervention will be determined acceptable if the overall median score is >= 4.
Time Frame: At 12 weeks
Population: Two participants did not complete this survey at 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Text Message Intervention
Number analyzed (Participants) | 44
score on a scale | 4 [3 to 4.5]

4. Primary Outcome: Overall Score on the Intervention Appropriateness Measure (IAM)
Description: The IAM is a four-item measure of implementation that assesses participants perceived appropriateness of the intervention. Each item response falls on a scale of 1 (Completely disagree) to 5 (Completely agree). A scaled score is calculated by averaging responses. Scale values range from 1 to 5. The intervention will be determined acceptable if the overall median score is >= 4.
Time Frame: At 12 weeks
Population: Two participants did not complete this survey at 12 weeks
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Text Message Intervention
Number analyzed (Participants) | 44
scores on a scale | 4 [3.4 to 4.9]

5. Primary Outcome: Feasibility of Intervention Measure (FIM)
Description: The FIM is a four-item measure of implementation that assesses participants perceived appropriateness of the intervention. Each item response falls on a scale of 1 (Completely disagree) to 5 (Completely agree). A scaled score is calculated by averaging responses. Scale values range from 1 to 5. The intervention will be determined acceptable if the overall median score is >= 4.
Time Frame: At 12 weeks
Population: Two participants did not complete this survey at 12 weeks
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Text Message Intervention
Number analyzed (Participants) | 44
scores on a scale | 4 [3.8 to 4]

6. Secondary Outcome: Change in Percent of Grains That Are Whole Reported on the Food Frequency Questionnaire (FFQ)
Description: The FFQ will ask about diet in the past 3 months. For each item, participants will be asked to report how often, on average, they ate the specified portion size in the past 3 months. Participants can choose from frequency options ranging from never or less than once per month to >=6 times a day. To compute calorie and nutrient intakes, multiply the frequency of consumption of each food by the amount of each nutrient in the specified portion size using composition values from the U.S. Department of Agriculture and other sources. Percent of grains that are whole = servings per day of whole grains/(servings per day of refined grains + servings per day of whole grains) will be reported over time
Time Frame: Up to 12 weeks
Population: Two participants did not complete this survey at 12 weeks
Measure: Median (95% Confidence Interval); unit: percentage of grains consumed
Arm/Group | Text Message Intervention
Number analyzed (Participants) | 44
percentage of grains consumed | 22.1 [13.5 to 30.7]

7. Secondary Outcome: Change in Mean Total Daily Fiber Intake (Grams Per Day (g/d)) Reported on the Food Frequency Questionnaire (FFQ)
Description: The FFQ will ask about diet in the past 3 months. For each item, participants will be asked to report how often, on average, they ate the specified portion size in the past 3 months. Participants can choose from frequency options ranging from never or less than once per month to >=6 times a day. To compute calorie and nutrient intakes, multiply the frequency of consumption of each food by the amount of each nutrient in the specified portion size using composition values from the U.S. Department of Agriculture and other sources. The mean total daily fiber intake and standard deviation will be reported over time.
Time Frame: Up to 12 weeks
Population: Two participants did not complete this survey at 12 weeks
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | Text Message Intervention
Number analyzed (Participants) | 44
grams per day | 4.3 (9.9)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: Pre-existing expected adverse events (e.g., diarrhea, constipation, etc.) were be assessed at enrollment and emergent events assessed at 12 weeks using a selected list of symptoms from the Patient reported outcome version of the CTCAE (PRO-CTCAE). Participants were also provided an opportunity to report additional symptoms not specifically selected in the PRO-CTCAE.
Arm/Group | Text Message Intervention
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 1/46
Other Adverse Events (participants affected / at risk) | 40/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Text Message Intervention (N=46)
Syncope (Fainted) (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Text Message Intervention (N=46)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Bloating (Gastrointestinal disorders) | 9 (9)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 8 (8)
Heartburn (Gastrointestinal disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (15)
Nausea (Gastrointestinal disorders) | 8 (8)
Paresthesia (Nervous system disorders) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT05746195/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT05746195/ICF_000.pdf